CLINICAL TRIAL: NCT04116853
Title: Evaluation of an Adaptive Intervention for Weight Loss Maintenance
Brief Title: Support and Tracking to Achieve Results (Project STAR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201803061 -N; R01DK119244 (NIH)
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-04

CONDITIONS: Obesity
Keywords: Weight Loss; Weight Maintenance
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: All randomized participants will receive extended-care intervention delivered via phone; however, the frequency/timing of these calls will vary between the ADAPTIVE and STATIC conditions.
Who Masked: Outcomes Assessor
Masking Description: Assessments will be conducted by trained study staff members masked to maintenance condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADAPTIVE Extended-Care Group (Experimental): Participants randomized to the ADAPTIVE extended-care program will receive extended-care intervention phone delivered only if either 1) an algorithm developed by our study team detects that a participant is at "high risk" for weight regain or 2) the participant self-initiates a request for a session.
  Interventions: Behavioral: ADAPTIVE Extended-Care Program
- STATIC Extended-Care Group (Active Comparator): Participants randomized to the STATIC extended-care program will receive the extended-care intervention phone calls on a fixed, once-per-month schedule (the schedule currently used in gold-standard weight maintenance programs).
  Interventions: Behavioral: STATIC Extended-Care Program

INTERVENTIONS:
Behavioral: ADAPTIVE Extended-Care Program — Each extended-care intervention phone call will be initiated by the interventionist, and will begin with a brief check-in followed by a discussion of any barriers experienced by participants in meeting their weight maintenance goals. Each call will end with a formal goal setting session. Calls are expected to last for approximately 10-20 minutes.
  Arms: ADAPTIVE Extended-Care Group
Behavioral: STATIC Extended-Care Program — Each extended-care intervention phone call will be initiated by the interventionist, and will begin with a brief check-in followed by a discussion of any barriers experienced by participants in meeting their weight maintenance goals. Each call will end with a formal goal setting session. Calls are expected to last for approximately 10-20 minutes.
  Arms: STATIC Extended-Care Group

SUMMARY:
The investigators propose to conduct a randomized controlled trial assessing the impact of phone-based extended care delivered on an ADAPTIVE (when participants are at "high risk" for weight regain as assessed by a predictive algorithm) vs. STATIC (gold-standard, once-per-month frequency) schedule on weight loss maintenance. The study team will provide participants with an initial behavioral weight management program, and then randomize participants who successfully achieve a clinically-significant weight loss of ≥5% to one of the two extended-care conditions

DETAILED DESCRIPTION:
Obesity remains a substantial public health challenge in the United States. While behavioral lifestyle interventions have been demonstrated to produce weight losses of 8-10% in adults with overweight and obesity, long-term outcomes are suboptimal, limiting effectiveness for long-term weight loss maintenance.

The study team will evaluate methods for providing phone-based extended-care to support weight loss maintenance. The investigators propose to conduct a randomized controlled trial assessing the impact of phone-based extended care delivered on an ADAPTIVE (when we determine that participants are at "high risk" for weight regain) vs. STATIC (once-per-month frequency used in gold-standard extended-care programs) schedule on weight loss maintenance. Participants will be provided with an initial in-person, group-based behavioral weight management program. Participants who successfully achieve a clinically-significant weight loss between baseline and Month 4 (defined by the Institute of Medicine as a reduction in weight of ≥ 5% from baseline) will be randomized into the clinical trial. Follow-up visits will occur at Month 12 and Month 24 after initial intervention baseline.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30.0-45.0 kg/m2
* Own a smartphone [Apple iPhone (5s or newer) or Android smartphone (KitKat OS 4.4 or newer)] with a cellular and data plan
* Weight ≤ 396 pounds (due to scale limit)
* Lose ≥ 5% of baseline weight during the initial weight loss intervention (Month 0 to Month 4)
* Completion of baseline assessment measures

Exclusion Criteria:

* History of bariatric surgery
* Current use of weight loss medications
* Weight loss of ≥ 10 lb in prior 6 months
* Physical limitations that prevent walking ¼ mile without stopping
* Use of a pacemaker
* Currently pregnant
* Currently breastfeeding
* Less than 1 year post-partum
* Plans to become pregnant within the study period
* Lack of written approval for participation from potential participant's physician if the participant has been diagnosed with type 2 diabetes, hypertension, or has a history of coronary heart disease
* More than one participant per household (enrollment limited to one participant per household)
* Medical conditions that contraindicate weight loss or prevent completion of the study (e.g., current diagnosis of cancer or terminal illness, dementia, or plans to relocate during the study period)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Ross, PhD, MPH, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ross KM, Swanson TN, Arroyo KM, Shetty A, Shankar MN, Krukowski RA. Within-week and within-year patterns in self-monitoring of dietary intake in adults with obesity participating in a behavioral weight loss program. Health Psychol Behav Med. 2025 Apr 2;13(1):2485476. doi: 10.1080/21642850.2025.2485476. eCollection 2025. PMID 40182625
- [Result] Shetty A, Ross KM. Associations Between Body Mass Index, Body Image Satisfaction, and Self-Weighing During a Behavioral Weight Loss Program. Obes Sci Pract. 2025 May 3;11(3):e70074. doi: 10.1002/osp4.70074. eCollection 2025 Jun. PMID 40321456
- [Result] Swanson TN, Bauman V, Ross KM. Associations between chronotype, weight loss, and adherence to caloric intake and physical activity goals during a behavioral weight loss intervention. J Behav Med. 2025 Aug;48(4):722-729. doi: 10.1007/s10865-025-00573-y. Epub 2025 May 7. PMID 40335844
- [Result] Ross KM, Carpenter CA, Arroyo KM, Shankar MN, Yi F, Qiu P, Anthony L, Ruiz J, Perri MG. Impact of transition from face-to-face to telehealth on behavioral obesity treatment during the COVID-19 pandemic. Obesity (Silver Spring). 2022 Apr;30(4):858-863. doi: 10.1002/oby.23383. Epub 2022 Mar 11. PMID 35037410
- [Result] Ross KM, Shankar MN, Qiu P, Tian Z, Ruiz J, Anthony L, Perri MG. Adaptive vs Monthly Support for Weight-Loss Maintenance: A Randomized Clinical Trial. JAMA Netw Open. 2025 Sep 2;8(9):e2532681. doi: 10.1001/jamanetworkopen.2025.32681. PMID 40982283
- [Result] Ross KM, Shankar MN, Qiu P, Tian Z, Swanson TN, Shetty A, Ruiz J, Anthony L, Perri MG. Design of Project STAR: A randomized controlled trial evaluating the impact of an adaptive intervention on long-term weight-loss maintenance. Contemp Clin Trials. 2024 Nov;146:107707. doi: 10.1016/j.cct.2024.107707. Epub 2024 Oct 9. PMID 39384066

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Adults with obesity were first offered a 16-week weight loss program; only participants who lost at least 5% of their baseline weight were eligible for randomization into the maintenance trial.
Period: Overall Study
Arm/Group | ADAPTIVE Extended-Care Group | STATIC Extended-Care Group
Started | 128 | 127
Month 12 | 126 | 120
Completed | 117 | 110
Not Completed | 11 | 17
Not completed — Adverse Event | 1 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Incarceration | 0 | 1
Not completed — Pregnancy | 1 | 1
Not completed — Began Other Weight Loss program | 4 | 8
Not completed — Began Anti-Obesity Medication | 3 | 3
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ADAPTIVE Extended-Care Group | STATIC Extended-Care Group | Total
Number analyzed (Participants) | 128 | 127 | 255
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (10.5) | 50.4 (12.1) | 50.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 99 | 209
  Male | 18 | 28 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 28 | 47
  White | 103 | 87 | 190
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 12 | 25
  Not Hispanic or Latino | 115 | 115 | 230
  Unknown or Not Reported | 0 | 0 | 0
Initial Weight Loss Program Weight Change [Mean (Standard Deviation); unit: % change] | -9.4 (3.3) | -9.6 (3.4) | -9.5 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Weight Change Month 4 to Month 24 of the ADAPTIVE Group Compared to the STATIC Group, Controlling for Initial Weight Loss
Description: Participant body weight will be measured at baseline, Month 4, Month 12, and Month 24 using study-provided BodyTrace e-scales. Participants will be asked to measure their weight first thing in the morning on a scheduled assessment day, before having anything to eat or drink but after using the restroom, in no more than light indoor clothing and with pockets emptied and shoes removed. Analyses will examine difference in weight change from Month 4 to 24 by group, controlling for initial weight loss (i.e., weight change from baseline to Month 4). Thus, although the outcome (weight) is assessed at each time point, the primary outcome is only a single comparison. Weight in kg at each time point are reported below (using intent-to-treat analyses, with multiple imputation used to handle missing data) along with the difference in weight change from Month 4 to Month 24 by group (Month 24 weight - Month 4 weight), controlling for initial weight loss (Month 4 weight - Baseline weight).
Time Frame: Baseline; Month 4; Month 12; Month 24
Population: These numbers differ from numbers reported under participant flow as we conducted intent-to-treat analyses, using all available data from all participant and multiple imputation used to handle missing data (see statistical analysis plan)
Measure: Mean (95% Confidence Interval); unit: Weight (kg)
Arm/Group | ADAPTIVE Extended-Care Group | STATIC Extended-Care Group
Number analyzed (Participants) | 128 | 127
Weight (kg)
  Baseline | 99.57 [97.12 to 102.02] | 100.22 [97.46 to 102.98]
  Month 4 | 90.18 [87.88 to 92.48] | 90.59 [87.85 to 93.33]
  Month 12 | 89.18 [86.73 to 91.63] | 90.15 [87.10 to 93.20]
  Month 24 | 91.45 [88.87 to 94.03] | 92.34 [89.26 to 95.42]
  Primary Outcome (weight change from Month 4 to 24, controlling for initial weight loss) | 1.27 [0.07 to 2.47] | 1.75 [0.43 to 3.06]

ADVERSE EVENTS:
Time Frame: From enrollment until the end of the study (Month 24)
Arm/Group | ADAPTIVE Extended-Care Group | STATIC Extended-Care Group
All-Cause Mortality (participants affected / at risk) | 0/128 | 1/127
Serious Adverse Events (participants affected / at risk) | 10/128 | 16/127
Other Adverse Events (participants affected / at risk) | 50/128 | 33/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADAPTIVE Extended-Care Group (N=128) | STATIC Extended-Care Group (N=127)
Autoimmune hemolytic anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Not related
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — Not related
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) — Not related
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Not related
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Not related
Dehydration (Gastrointestinal disorders) | 0 (0) | 2 (2) — (vomiting / diarrhea)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Nerve damage in arm and neck after car accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headaches and tinnitus (Investigations) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Seizure after car accident (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Gallbladder removal (Surgical and medical procedures) | 1 (1) | 2 (2)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Hernia surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Shoulder replacement surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Heart bypass surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
C5 and C6 vertebrae surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Neurosurgery for Chiari malformation (Surgical and medical procedures) | 0 (0) | 1 (1)
Laparoscopic cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADAPTIVE Extended-Care Group (N=128) | STATIC Extended-Care Group (N=127)
COVID-19 (Infections and infestations) | 17 (17) | 9 (9)
Sinusitis (Infections and infestations) | 6 (6) | 7 (7)
Trip/Fall (Injury, poisoning and procedural complications) | 10 (10) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 8 (9)
Tooth extraction (Surgical and medical procedures) | 10 (10) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT04116853/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT04116853/ICF_001.pdf